CLINICAL TRIAL: NCT02320266
Title: Sensory Gating Measured With Microelectrode Recording During Deep Brain Stimulation Surgery
Brief Title: Sensory Gating Measured With Microelectrode Recording (MER) During Deep Brain Stimulation (DBS) Surgery
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0358
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Parkinson's Disease; Essential Tremor; Dystonia; Obsessive Compulsive Disorder
Keywords: Deep Brain Stimulation Surgery
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Dystonia; Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Parkinson's Disease: Patients diagnosed with Parkinson's Disease undergoing DBS surgery.
- Control: Age matched controls without Parkinson's Disease and no history of mental illness.
- Essential Tremor: Patients diagnosed with Essential Tremor undergoing DBS surgery.
- Dystonia: Patients diagnosed with Dystonia undergoing DBS surgery.
- Obsessive-Compulsive disorder: Patients diagnosed with Obsessive-Compulsive disorder undergoing DBS surgery.

SUMMARY:
Deep brain stimulation (DBS) is an FDA approved, and widely used method for treating the motor symptoms of Parkinson's disease (PD), Essential Tremor (ET), Dystonia and Obsessive Compulsive disorder (OCD). Over 100,000 patients worldwide have now been implanted with DBS devices. Current approved methods to locate the DBS target regions in the brain use a combination of stereotactic imaging techniques and measurements of the electrical activity of brain cells. As part of the standard clinical technique, electrical data are collected from individual nerve cells. The target brain region emits unique electrical signals. At certain brain locations, during DBS surgery, additional electrical data that are generated in response to sound will be collected. Regions of the brain that have a decreased response to repeated sound (auditory gating) may be important DBS targets for improving thinking. The aims are (i) during DBS surgery, in addition to EEG, use microelectrodes in the brain to find brain regions, along the normal path to the DBS target, where auditory gating occurs and then (ii) determine if stimulation of the identified region(s) alters auditory gating measured by EEG. Also an additional aim (iii) is to measure electrical activity at the scalp with EEG to characterize auditory gating in patients before and after DBS surgery and also a healthy control population.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) is an FDA approved, and widely used method for treating the motor symptoms of Parkinson's disease (PD), Essential Tremor (ET), Dystonia and Obsessive Compulsive disorder (OCD). Over 100,000 patients worldwide have now been implanted with DBS devices. Current approved methods to locate the DBS target regions in the brain (subthalamic nucleus (STN) for PD) use a combination of stereotactic imaging techniques and measurements of the electrical activity of brain cells. As part of the standard clinical technique, electrical data are collected from individual nerve cells --in a procedure called microelectrode recording (MER). The target brain region emits unique electrical signals that are detected by MER during the standard DBS surgery. MER is done at stops along the way to the target. At the stops during DBS surgery, additional electrical data that are generated in response to sound will be collected. Regions of the brain that have a decreased response after repeated sound (auditory gating) may be important DBS targets for improving thinking. The aims are to:(Aim 1A) during DBS surgery, in addition to EEG, use microelectrodes in the brain to measure electrical activity with single unit activity (SUA) and local field potentials (LFP) to find brain regions along the path to the DBS target where auditory gating occurs (Aim 1A) and then determine if stimulation of the identified region(s) alters auditory gating measured by EEG(Aim 1B); and (Aim 2) measure electrical activity at the scalp with electroencephalography (EEG) to characterize auditory gating in patients before and after DBS surgery and also a healthy control population.

ELIGIBILITY:
Inclusion Criteria:

* subjects with Parkinson's Disease planning to undergo DBS surgery
* subjects without Parkinson's Disease
* subjects without a history of mental illness.

Exclusion Criteria:

* subjects with hearing impairment
* illicit drug use
* marijuana use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with Parkinson's Disease who are planning to undergo DBS surgery. Age matched controls without Parkinson's Disease or a history of mental illness.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-12; Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in EEG (Measurement in response to paired auditory clicks.) | 20 min to 2 hours
  Measurement in response to paired auditory clicks.
Evaluation of SUA (Single unit analysis of brain response.) | 20 min
  Single unit analysis of brain response.
Evaluation of LFP (Local field potential of brain response.) | 20 min
  Local field potential of brain response.

CONTACTS AND LOCATIONS:
Overall Officials: Judith M Gault, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States